CLINICAL TRIAL: NCT06903416
Title: Comparative Evaluation of Non-Invasive Neuromodulation Therapies to Restore Upper Extremity Function in Chronic Cervical Spinal Cord Injury
Brief Title: Non-Invasive Neuromodulation for Upper Extremity Function in Spinal Cord Injury: A Crossover Trial
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Praxis Spinal Cord Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00149698
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury Cervical

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Transcutaneous Spinal Cord Stimulation with Functional Task Practice (Active Comparator): Cervical transcutaneous spinal cord stimulation will be delivered following previously reported guidelines. Circular (1.25") electrodes will be placed over the cervical spinal cord between the C3 and C4 vertebral level, with rectangular return electrodes placed either over the clavicles or iliac crests. Biphasic stimulation will be delivered continuously at 30Hz, with a 1ms pulse width, and overlapping 10kHz carrier frequency (Gelenitis et al 2024; Moritz et al 2024). Stimulation will be delivered at a current intensity below motor threshold, that is below the intensity required to elicit a muscle twitch. Cervical tSCS will be delivered for at least 60 minutes during each training session, and FTP will occur during the active stimulation.
  Interventions: Other: Transcutaneous Cervical Spinal Cord Stimulation; Other: Functional Task Practice
- Paired Corticospinal Motoneuronal Stimulation with Functional Task Practice (Active Comparator): Paired transcranial magnetic stimulation and nerve stimulation will be implemented following a previously-published protocol for individuals with SCI (Jo et al 2023). Two figure-eight coils will be used to deliver bilateral magnetic stimulation of the motor cortex and will be combined with synchronous electrical stimulation of the brachial plexus and ulnar nerves, bilaterally. The timing of stimuli will be determined to ensure that electrical volleys arrive at the corticospinal motoneuronal synapse at an appropriate interval to induce long term potentiation. During each session, 360 paired stimuli will be delivered at a frequency of 0.2 Hz. The stimulation paradigm should take approximately 30 minutes. Following this, participants will then complete 60 minutes of FTP.
  Interventions: Other: Paired Corticospinal Motoneuronal Stimulation; Other: Functional Task Practice

INTERVENTIONS:
Other: Transcutaneous Cervical Spinal Cord Stimulation — Cervical transcutaneous spinal cord stimulation will be delivered following previously reported guidelines. Circular (1.25") electrodes will be placed over the cervical spinal cord between the C3 and C4 vertebral level, with rectangular return electrodes placed either over the clavicles or iliac crests. Biphasic stimulation will be delivered continuously at 30Hz, with a 1ms pulse width, and overlapping 10kHz carrier frequency (Gelenitis et al 2024; Moritz et al 2024). Stimulation will be delivered at a current intensity below motor threshold, that is below the intensity required to elicit a muscle twitch. Cervical tSCS will be delivered for at least 60 minutes during each training session, and FTP will occur during the active stimulation.
  Arms: Cervical Transcutaneous Spinal Cord Stimulation with Functional Task Practice
Other: Paired Corticospinal Motoneuronal Stimulation — Paired transcranial magnetic stimulation and nerve stimulation will be implemented following a previously-published protocol for individuals with SCI (Jo et al 2023). Two figure-eight coils will be used to deliver bilateral magnetic stimulation of the motor cortex and will be combined with synchronous electrical stimulation of the brachial plexus and ulnar nerves, bilaterally. The timing of stimuli will be determined to ensure that electrical volleys arrive at the corticospinal motoneuronal synapse at an appropriate interval to induce long term potentiation. During each session, 360 paired stimuli will be delivered at a frequency of 0.2 Hz. The stimulation paradigm should take approximately 30 minutes. Following this, participants will then complete 60 minutes of FTP.
  Arms: Paired Corticospinal Motoneuronal Stimulation with Functional Task Practice
Other: Functional Task Practice — A typical rehabilitation program will be defined and delivered in consultation with physical and occupational therapists. The program will consist of functional tasks including repetitive activities of gross upper extremity movement, isolated finger movements, simple and complex pinch, and grasping activities. For each category, 4-10 activities with various difficulty levels will be identified. Each participant will perform at least 1-2 exercises within each category during each treatment session. Activities in each category will be chosen according to the participants' ability and adjusted based on the evolution of the ability to perform the functional task over time (graded training).

SUMMARY:
This study explores two promising therapies for restoring arm and hand function in people with chronic cervical spinal cord injury (SCI), a condition that affects independence and quality of life. It will compare transcutaneous spinal cord stimulation and paired corticospinal-motoneuronal stimulation, both combined with rehabilitation. Using a crossover design, participants will receive each therapy for two months, with a one-month washout period in between. Safety, effectiveness, and patient-reported outcomes like daily living ability and quality of life will be assessed, alongside changes in neural excitability. The results of this study may enable us to tailor treatments to individual needs, promoting personalized care and improved outcomes.

DETAILED DESCRIPTION:
Project Aims

The key objective of this pilot is to explore the feasibility of a comparative trial between two non-invasive neuromodulatory approaches for restoration of upper extremity function after SCI, and to work towards the identification of participant cohorts most suited for each intervention (i.e. responders). This objective will be achieved through the following:

1. Evaluation of clinical safety and effectiveness of each intervention, within participants, through safety monitoring and the use of standardized assessments of upper extremity strength, sensation and movement performance.
2. Evaluation of clinically meaningful improvements through participant reported outcomes related to activities of daily living, QoL and global impressions of change.
3. Neurophysiological assessments to assess the mechanisms of recovery following each interventional period, but also to aid in the identification of neurophysiological correlates of "responders" to each therapy.

In this randomized crossover study, participants will receive two months of non-invasive tSCS over the cervical spinal cord in combination with functional task practice (minimum of 12 sessions/month) preceded or followed by two months of PCMS and functional task practice, with a 4-week washout period between each intervention. With this design we will be able to examine the relative efficacy of each paradigm within a single participant and begin to identify neurophysiological and/or clinical characteristics that may help to guide the clinical identification of suitable participants for each intervention.

The minimum training dose for each interventional block is 12 sessions/month, for a total of 24 sessions of training during each treatment phase. Participants will be invited to complete up to 5 sessions per week if feasible. Participants will be required to complete a comparable number of intervention sessions (i.e., within 10%) in each of the two interventions to ensure that any effects are not attributed to differences in dosage. Each intervention session will include at least 60 minutes of upper extremity functional task practice (FTP). The FTP will be completed with typical rehabilitation activities (e.g., range of motion, strengthening activities, moving paperclips, clothespins, cups, etc.) as well as the ReJoyce rehabilitation workstation (Rehabtronics, Alberta), which incorporates computer games into the rehabilitation activities.

Transcutaneous Cervical Spinal Cord Stimulation (tSCS) Cervical transcutaneous spinal cord stimulation will be delivered following previously reported guidelines. Circular (1.25") electrodes will be placed over the cervical spinal cord between the C3 and C4 vertebral level, with rectangular return electrodes placed either over the clavicles or iliac crests. Biphasic stimulation will be delivered continuously at 30Hz, with a 1ms pulse width, and overlapping 10kHz carrier frequency (Gelenitis et al 2024; Moritz et al 2024). Stimulation will be delivered at a current intensity below motor threshold, that is below the intensity required to elicit a muscle twitch. Cervical tSCS will be delivered for at least 60 minutes during each training session, and FTP will occur during the active stimulation.

Paired Corticospinal Motoneuronal Stimulation (PCMS) Paired transcranial magnetic stimulation and nerve stimulation will be implemented following a previously-published protocol for individuals with SCI (Jo et al 2023). Two figure-eight coils will be used to deliver bilateral magnetic stimulation of the motor cortex and will be combined with synchronous electrical stimulation of the brachial plexus and ulnar nerves, bilaterally. The timing of stimuli will be determined to ensure that electrical volleys arrive at the corticospinal motoneuronal synapse at an appropriate interval to induce long term potentiation. During each session, 360 paired stimuli will be delivered at a frequency of 0.2 Hz. The stimulation paradigm should take approximately 30 minutes. Following this, participants will then complete 60 minutes of FTP.

Functional Task Practice (FTP) A typical rehabilitation program will be defined and delivered in consultation with physical and occupational therapists. The program will consist of functional tasks including repetitive activities of gross upper extremity movement, isolated finger movements, simple and complex pinch, and grasping activities. For each category, 4-10 activities with various difficulty levels will be identified. Each participant will perform at least 1-2 exercises within each category during each treatment session. Activities in each category will be chosen according to the participants' ability and adjusted based on the evolution of the ability to perform the functional task over time (graded training).

Assessment Measures

Assessments will occur at baseline then monthly for five months, corresponding to the beginning, midpoint and end of each treatment block. All participants will also have a three-month follow-up assessment to evaluate retention of any intervention effects (i.e. carryover neuroplasticity).

Outcomes Clinical measures will be completed by an occupational or physical therapist who is blinded to participants' group allocation. Assessments will include clinical measures of upper extremity strength, sensation and function including the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) and related subscores such as Upper Extremity Motor Score and Sensory Scores as well as the Graded Redefined Assessment of Strength Sensation and Performance (GRASSP). Patient reported outcomes will evaluate self-reported ability to perform activities of daily living (SCIM-III), overall quality of life (WHO-QoL BREF) and participant global impressions of change (PGIC) at the beginning and end of each intervention block (Figure 1).

Neurophysiological assessments will include transcranial magnetic stimulation (TMS) over the upper limb motor cortex to assess the excitability of the corticospinal tract, as well as stimulation to cervical dorsal roots to evaluate changes in cervical spinal cord excitability from the evoked multisegmental motor responses (cMMRs). TMS of the cortex has been used extensively in humans to assess the integrity of the descending corticospinal tract (Di Lazzaro et al 2008). Participants will be seated in their wheelchair. Single pulse TMS will be delivered at increasing stimulation intensity, with three stimuli (5s apart) at each intensity, until a plateau in evoked responses is reached, or we reach 100% maximal stimulator output or participant tolerability. Surface EMG will be recorded from multiple upper extremity muscles, bilaterally.

In a single visit, cMMRs will be evoked transcutaneously using single stimuli (1ms monophasic pulse). Muscle responses will be collected from multiple upper extremity muscles as per above. Stimulation will be delivered at an intensity below motor threshold for all muscles and will then be increased progressively until a plateau in evoked responses across the multiple muscles is obtained, or until participant tolerance is reached. The intensity increments will be chosen to ensure at least 9 measurements along the linear portion of the recruitment curve. Participants will receive 3 stimuli at each intensity, and stimuli will be delivered 5s apart (D'Amico et al 2013). Maximal compound muscle action potentials (Mmax) will be obtained at completion of the session by supramaximal stimulation of the brachial plexus (0.2ms pulse width).

Data Analysis Neurophysiology Measures The area of the reflex responses and MEPs obtained from TMS will be normalized to the Mmax area corresponding to the same muscle. The areas (%Mmax) will be plotted against the stimulation intensity (as a % maximum stimulator output (%MSO) or % of motor threshold (xMT)) and fit with a 3-parameter sigmoid function (D'Amico et al 2020, Klimstra & Zehr 2008). The stimulation intensity required to elicit a response 50% of the maximum response (S50) and the maximum evoked responses (cMMRmax) will be calculated for each muscle by fitting the experimental data with a three-parameter sigmoid function (D'Amico et al 2013, Klimstra & Zehr 2008). These measures will then be compared between the two interventions (tSCS and PCMS) within each participant.

Clinical and Patient-Reported Outcome Measures Scores on each patient-reported outcome measure and clinical assessment will follow the standard protocol for scoring each assessment. All scores will be compared between baselines, end of each intervention period, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Cervical (C2-C8) level SCI
* > 9 months post-injury
* Traumatic SCI
* AIS A-D
* Stable dose of anti-spasmodics

Exclusion Criteria:

* individuals with injury to the nervous system other than to the spinal cord
* pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2030-03-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | Baseline, 2 months (end of block 1), 3 months (start of block 2), 5months (end of block 2) and 8 months (follow-up)
  The ISNCSCI and its associated subscores related to upper extremity motor and sensory scores will be completed by a blinded assessor.
Graded Redefined Assessment of Strength Sensation and Performance (GRASSP) | Baseline, 2 months (end of block 1), 3 months (start of block 2), 5months (end of block 2) and 8 months (follow-up)
  The GRASSP will be assessed by a blinded assessor to evaluate changes in strength, sensation and performance of the upper extremities.

SECONDARY OUTCOMES:
Spinal excitability - Cervical Multisegmental Motor Responses (cMMR) | Baseline, 1 month (mid-block 1), 2 months (end of block 1), 3 months (start of block 2), 4 months (mid block 2), 5months (end of block 2) and 8 months (follow-up)
  Electrical stimulation to cervical dorsal roots via electrodes placed over the midline of the spinal cord will be used to evaluate changes in cervical spinal cord excitability from the intervention. Recruitment curves will be performed by progressively increasing the stimulation intensity until a plateau in evoked response or reached, or until participant tolerance is reached.
Corticospinal Excitability-Transcranial magnetic stimulation (TMS) | Baseline, 1 month (mid-block 1), 2 months (end of block 1), 3 months (start of block 2), 4 months (mid block 2), 5months (end of block 2) and 8 months (follow-up)
  TMS of the cortex has been used extensively in humans to assess the integrity of the descending corticospinal tract (Di Lazzaro et al 2008). Participants will be seated in their wheelchair. Single pulse TMS will be delivered at increasing stimulation intensity, with three stimuli (5s apart) at each intensity, until a plateau in evoked responses is reached, or we reach 100% maximal stimulator output or participant tolerability. Surface EMG will be recorded from multiple upper extremity muscles, bilaterally.

OTHER OUTCOMES:
SCIM III | Baseline, 2 months (end of block 1), 3 months (start of block 2), 5months (end of block 2) and 8 months (follow-up)
  The SCIM III is a validated survey for people with SCI that assesses independence during activities of daily living such as self-care, respiration and sphincter management and mobility. Participants will complete this survey themselves.
WHOQoL-BREF | Baseline, 2 months (end of block 1), 3 months (start of block 2), 5months (end of block 2) and 8 months (follow-up)
  The WHOQoL-BREF will be self-reported by participants to assess changes in the four domains: physical, psychological, social and environment.
Patient Global Impression of Change (PGIC) Score | Month 2 (end of block 1), and Month 5 (end of block 2)
  Participant will self-report their impressions of change upon completion of each phase of the interventional crossover study.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M D'Amico, PhD, Principal Investigator — University of Alberta
Locations (1):
- Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan to shared IPD with other researchers. Deidentified data may be shared with a data repository.